CLINICAL TRIAL: NCT00582842
Title: Longitudinal Assessment of Health-Related Quality of Life in Men With Localized Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 02-042
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
Keywords: Early Stage; Localized
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Men with prostate cancer
  Interventions: Behavioral: Interview
- 2: Men with prostate cancer
  Interventions: Behavioral: survey instruments using Web-Based Data Collection System (WBDC) survey content

INTERVENTIONS:
Behavioral: Interview — The phone interview will consist of the following items from the follow up questionnaire; 14, 16, 20, 32, 33, 46, 47, 60, and 65. An additional component of this study would be dispensing the HRQOL tool to long-term survivors 10 years or greater after the completion of therapy. The long term QoL study will be a cross-sectional assessment measuring HRQOL in prostate cancer survivors, free of disease at least ten years post-treatment. Patients will complete a questionnaire by selfreport focusing on assessment of HRQOL.
  Groups: 1
Behavioral: survey instruments using Web-Based Data Collection System (WBDC) survey content — The content of the WBDC questionnaire will be similar to the paper form, no alteration in the wording, the order, or the formate of the items will be done. In addition, at the time of each outpatient clinic visit to MSKCC, these subjects will be able to login to WBDC using a computer located in the patient waiting-area, and enter their responses to the different items of the questionnaire if their clinic visit corresponds to any of the study time points 3, 6, 9, 12, 15, 18, 24, 36, and 48 following treatment). An additional component of this study would be dispensing the HRQOL tool to long-term survivors 10 years or greater after the completion of therapy. The long term QoL study will be a cross-sectional assessment measuring HRQOL in prostate cancer survivors, free of disease at least ten years post-treatment. Patients will complete a questionnaire by selfreport focusing on assessment of HRQOL.
  Groups: 2

SUMMARY:
The purpose of this study is to assess quality-of-life of men with prostate cancer. "Quality-of-life" means how you feel about your life as a result of your disease and its treatment. The investigators hope that this questionnaire will help show how prostate cancer treatments affect quality-of-life. It will help doctors and future patients to make better treatment choices. Some men may wish to have a more demanding treatment with a higher risk of harmful effects. Others may prefer a treatment that will have the smallest effect on their quality-of-life.

This questionnaire will help us measure these effects and decide which is the best treatment for a given patient.

DETAILED DESCRIPTION:
The intent of the protocol is to assess health-related quality-of-life (HRQOL) in men treated for localized prostate cancer with 1 of 6 established management alternatives: external (XRT)or interstitial radiotherapy (IRT), open radical prostatectomy (RP), laparoscopic radical prostatectomy (LRP), combined radiotherapy and brachytherapy (Combined RT) or watchful waiting (WW). HRQOL is an important aspect of any treatment for prostate cancer due to the beliefs by many that cancer control rates are similar across common modalities and HRQOL reduction from treatment is substantial (1-5). Therefore, HRQOL appears to occupy a central role in the decision making process related to treatment selection.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of localized, untreated prostate cancer (clinical stages T1-3, Nx, M0)
* ability to read the English language

Exclusion criteria:

* other cancer diagnosis for the past three years, except for non-melanoma skin cancer
* prior chemotherapy within the last three years; radiation therapy to the pelvis or prior pelvic surgery within the past three years
* prior neoadjuvant therapy, such as hormones (Bicalutamide use for less than or equal to 1 month would not constitute exclusion from study entry)

For the cross-sectional component of the study, all patients identified to be free of disease at least ten years post -treatment will be considered eligible. Patients must have no clinical evidence of local, regional or distant recurrences. Patients must have the ability to read and understand English. Patients who received hormonal therapy will be eligible for the cross-sectional component of the study, but the duration of the hormonal therapy must be six months or less. the investigators have identified a cohort of patients who fit these criteria from our databases.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible MSKCC patients (including patients from the regional network sites: Commack, Basking Ridge, Rockville Centre and Sleepy Hollow) will be approached by consenting professionals and invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2002-05-14 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Assessment of temporal trends in HRQOL according to intervention group | study time points 3, 6, 9, 12, 15, 18, 24, 36, and 48 following treatment)and between 60 and 96 months.

SECONDARY OUTCOMES:
Assessment of scale score differences between treatment groups | 3, 6, 9, 12, 15, 18, 24, 36, 48 months and between 60 and 96 months
Describe the quality of life of long-term survivors | 10 years post treatment
  of prostate cancer following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Scardino, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer website — http://www.mskcc.org